CLINICAL TRIAL: NCT02256722
Title: A Randomised, Open Label, Four-way Crossover Phase I Trial to Investigate the in Vivo Specificity of a Single Oral Dose of 320 mg KUC 7483 CL Co-administered With Bisoprolol (10 mg Daily), Propranolol (160 mg Daily), and Acipimox (500 mg Daily) Over 5 Days and a Single Inhalative Dose of 100 μg Salmeterol in Healthy Male Subjects
Brief Title: In Vivo Specificity of KUC 7483 CL Co-administered With Bisoprolol, Propranolol, and Acipimox in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1207.26
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Bisoprolol; Propranolol; acipimox; Salmeterol Xinafoate

ARMS (5):
- Treatment A (Experimental)
  Interventions: Drug: KUC 7483 CL
- Treatment B (Experimental)
  Interventions: Drug: KUC 7483 CL; Drug: Bisoprolol
- Treatment C (Experimental)
  Interventions: Drug: KUC 7483 CL; Drug: Propranolol
- Treatment D (Experimental)
  Interventions: Drug: KUC 7483 CL; Drug: Acipimox
- Treatment E (Active Comparator)
  Interventions: Drug: Salmeterol

INTERVENTIONS:
Drug: KUC 7483 CL
  Arms: Treatment A; Treatment B; Treatment C; Treatment D
Drug: Bisoprolol
  Arms: Treatment B
Drug: Propranolol
  Arms: Treatment C
Drug: Acipimox
  Arms: Treatment D
Drug: Salmeterol
  Arms: Treatment E

SUMMARY:
Study to compare the metabolic and electrolyte effects of a single oral dose of 320 mg ritobegron administered alone or with a pre- and comedication with bisoprolol, propranolol and acipimox. In addition, to compare the metabolic and electrolyte effects of a single dose of 320 mg ritobegron with those of a single inhalatory dose of 100 μg salmeterol

ELIGIBILITY:
Inclusion Criteria:

* Healthy male
* Age >= 30 and <= 60 years
* Body Mass Index (BMI) >= 18.5 and <= 29.9 kg/m2
* Signed and dated written informed consent in accordance with Good Clinical Practice and local legislation

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders, clinically relevant electrolyte disturbances
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or clinically relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24:00 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study or during the study
* Use of any drugs which might influence the results of the trial up to 7 days prior to enrolment in the study or during the study
* Participation in another trial with an investigational drug (within two months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars of > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (> 100 mL within four weeks prior to administration or during the trial)
* Any laboratory value outside the reference range if indicative of underlying disease or poor health
* Excessive physical activities within the last week before the trial or during the trial
* Hypersensitivity to treatment medication, salmeterol and/or related drugs of these classes
* Congenital or documented acquired QT- prolongation, previous history of symptomatic arrhythmias
* Systolic BP < 115 mmHg
* Heart rate at rest of > 80 bpm or < 55 bpm
* Any screening ECG value outside of the reference range of clinical relevance including, but not limited to PR interval > 220 ms, QRS interval > 115 ms, QTcB > 420 ms, or QT (uncorrected) > 450 ms
* History of asthma or obstructive pulmonary disease.
* Psoriasis (own medical history or relative)

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2005-10; Primary Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline in glucose | up to 24 hours after administration of study drug
Percentage change from baseline in glucose | up to 24 hours after administration of study drug
Absolute change from baseline in free fatty acids (FFA) | up to 24 hours after administration of study drug
Percentage change from baseline in FFA | up to 24 hours after administration of study drug
Absolute change from baseline in insulin | up to 24 hours after administration of study drug
Percentage change from baseline in insulin | up to 24 hours after administration of study drug
Absolute change from baseline in C-Peptide | up to 24 hours after administration of study drug
Percentage change from baseline in C-Peptide | up to 24 hours after administration of study drug
Absolute change from baseline in Potassium | up to 24 hours after administration of study drug
Percentage change from baseline in Potassium | up to 24 hours after administration of study drug
Absolute change from baseline in Magnesium | up to 24 hours after administration of study drug
Percentage change from baseline in Magnesium | up to 24 hours after administration of study drug
Absolute change from baseline in cAMP | up to 24 hours after administration of study drug
Percentage change from baseline in cAMP | up to 24 hours after administration of study drug

SECONDARY OUTCOMES:
Number of subjects with adverse events | up to 80 days
Number of subjects with clinically relevant changes in laboratory tests | up to 24 hours after administration of study drug
Number of subjects with clinically relevant changes in vital signs | up to 24 hours after administration of study drug
Number of subjects with clinically relevant findings in electrocardiogram | up to 24 hours after administration of study drug
Number of subjects with clinically relevant changes in physical examination | Baseline, within 10 days after last drug administration
Maximum measured concentration of the analyte in plasma | up to 24 hours after administration of study drug
Time from dosing to the maximum concentration of the analyte in plasma | up to 24 hours after administration of study drug
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 4 hours | up to 24 hours after administration of study drug